CLINICAL TRIAL: NCT02813044
Title: Effects of Total Intravenous Anesthesia With Propofol-remifentanil Versus Inhalational Anesthesia With Sevoflurane on Quality of Recovery in Patients Undergoing Transsphenoidal Surgery for Pituitary Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2016-0344
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Pituitary Tumor
Keywords: anesthesia; intravenous; neurosurgery; pituitary neoplasm; postoperative period
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIVA group (Experimental): Anesthesia is maintained with propofol during surgery
  Interventions: Drug: total intravenous anesthesia (TIVA)
- inhalation anesthesia group (Active Comparator): Anesthesia is maintained with sevoflurane during surgery
  Interventions: Drug: inhalation anesthesia group

INTERVENTIONS:
Drug: total intravenous anesthesia (TIVA) — In the TIVA group,anesthesia is induced and maintained by effect-site target controlled infusion of propofol and remifentanil.
  Arms: TIVA group
Drug: inhalation anesthesia group — In the inhalation anesthesia group, anesthesia is induced by pentothal sodium 4-6mg/kg and remifentanil 1 μg/kg, and then maintained with end-tidal sevoflurane concentration of 0.8 to 1 MAC and continuous infusion of remifentanil at 0.1-0.3μg/kg/min.
  Arms: inhalation anesthesia group

SUMMARY:
A number of studies have compared the effects of total intravenous anesthesia(TIVA) versus inhalational anesthesia on perioperative period during transsphenoidal surgery. However, they have limitations especially for the phase of recovery after anesthesia: a fragmentary assessment. Quality of Recovery 40 (QoR-40) questionnaire was multi-dimensionally designed to assess the degree of recovery, specially after anesthesia and surgery. In this study, the investigators aim to compare the quality of recovery after inhalational anesthesia and after TIVA through QoR-40 questionnaire in patients undergoing transsphenoidal surgery for pituitary tumor under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over age 19
* Scheduled to undergo transsphenoidal surgery for pituitary tumor
* ASA class I and II

Exclusion Criteria:

* Left ventricular ejection fraction < 55%
* Third-degree atrioventricular block
* Second-degree atrioventricular block (P:QRS ratio of 3:1 or higher)
* Fever
* History of myocardial infarction, stroke or cardiac surgery within the previous 1 year
* Severe neurological disease
* Use of sedative, opioid or sleep-inducing drugs
* Allergic history of any study drug
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
QoR-40 score | 1 day
  We compare the QoR-40 scores of two groups 1 day after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Associate Professor Department of Anesthesiology and Pain Medicine,, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Shaikh B, George William M, Van Zundert AA. Using atmospheric pressure to inflate the cuff of the Portex Laryngeal Mask. Anaesthesia. 2005 Mar;60(3):296-7. doi: 10.1111/j.1365-2044.2005.04135.x. No abstract available. PMID 15710025